CLINICAL TRIAL: NCT06673641
Title: A Multi-center, Double-blind, Randomized, Placebo-controlled, Parallel-group Study, Comparing Clindamycin Phosphate, Adapalene, and Benzoyl Peroxide Topical Gel 0.15%;3.1%;1.2% to CABTREO (Clindamycin Phosphate, Adapalene, and Benzoyl Peroxide) Topical Gel and Both Active Treatments to a Placebo Control in the Treatment of Acne Vulgaris.
Brief Title: A Study Comparing Clindamycin Phosphate, Adapalene, and Benzoyl Peroxide Topical Gel 0.15%;3.1%;1.2% (Taro Pharmaceuticals U.S.A., Inc.) and CABTREO Topical Gel for the Treatment of Acne Vulgaris.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sun Pharmaceutical Industries, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ABCG-2407
Record Dates: First submitted 2024-11-02; First posted 2024-11-05 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-10

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — clindamycin phosphate; Adapalene

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Clindamycin Phosphate, Adapalene, and Benzoyl Peroxide Topical Gel 0.15%;3.1%;1.2% (Experimental): The study medication was applied once daily to cover the entire face after washing, avoiding the eyes, lips, angles of the nose, and mucous membranes for 84 consecutive days.
  Interventions: Drug: Clindamycin Phosphate, Adapalene, and Benzoyl Peroxide Topical Gel 0.15%;3.1%;1.2%
- CABTREO Topical Gel (Active Comparator): The study medication was applied once daily to cover the entire face after washing, avoiding the eyes, lips, angles of the nose, and mucous membranes for 84 consecutive days.
  Interventions: Drug: CABTREO Topical Gel
- Placebo Control (Placebo Comparator): The study medication was applied once daily to cover the entire face after washing, avoiding the eyes, lips, angles of the nose, and mucous membranes for 84 consecutive days.
  Interventions: Drug: Placebo Control

INTERVENTIONS:
Drug: Clindamycin Phosphate, Adapalene, and Benzoyl Peroxide Topical Gel 0.15%;3.1%;1.2% — The study medication was applied once daily to cover the entire face after washing, avoiding the eyes, lips, angles of the nose, and mucous membranes for 84 consecutive days.
  Other Names: Test Product
  Arms: Clindamycin Phosphate, Adapalene, and Benzoyl Peroxide Topical Gel 0.15%;3.1%;1.2%
Drug: CABTREO Topical Gel — The study medication was applied once daily to cover the entire face after washing, avoiding the eyes, lips, angles of the nose, and mucous membranes for 84 consecutive days.
  Other Names: Reference Product
  Arms: CABTREO Topical Gel
Drug: Placebo Control — The study medication was applied once daily to cover the entire face after washing, avoiding the eyes, lips, angles of the nose, and mucous membranes for 84 consecutive days.
  Other Names: Vehicle
  Arms: Placebo Control

SUMMARY:
To demonstrate the efficacy, therapeutic equivalence and safety of Clindamycin Phosphate, Adapalene, and Benzoyl Peroxide Topical Gel 0.15%;3.1%;1.2% (Taro Pharmaceuticals U.S.A., Inc.) and CABTREO Topical Gel in the treatment of acne vulgaris.

DETAILED DESCRIPTION:
A multi-center, double-blind, randomized, placebo-controlled, parallel-group study, comparing Clindamycin Phosphate, Adapalene, and Benzoyl Peroxide topical gel 0.15%;3.1%;1.2% to CABTREO (Clindamycin Phosphate, Adapalene, And Benzoyl Peroxide) topical gel in the treatment of acne vulgaris.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or nonpregnant female aged ≥ 12 and ≤ 40years with a clinical diagnosis of acne vulgaris.
* Subjects who are 18 years of age or older must have provided IRB approved written informed consent.
* Subjects must have a definite clinical diagnosis of acne vulgaris severity grade 2, 3 or 4 as per the Investigator's Global Assessment (IGA).
* Subjects must have ≥ 25 non-inflammatory lesions (i.e., open and closed comedones) AND ≥ 20 inflammatory lesions (i.e., papules and pustules) AND ≤2 nodulocystic lesions (i.e., nodules and cysts), at baseline on the face.

Exclusion Criteria:

* Female Subjects who are pregnant, nursing or planning to become pregnant during study participation.
* Subjects with a history of hypersensitivity or allergy to clindamycin phosphate, benzoyl peroxide, adapalene, retinoids and/or any of the study medication ingredients.
* Subjects with the presence of any skin condition that would interfere with the diagnosis or assessment of acne vulgaris (e.g., on the face: rosacea, dermatitis, psoriasis, squamous cell carcinoma, eczema, acneiform eruptions caused by medications, steroid acne, steroid folliculitis, or bacterial folliculitis).
* Subjects with excessive facial hair (e.g. beards, sideburns, mustaches, etc.) that would interfere with the diagnosis or assessment of acne vulgaris.

Ages: 12 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 382 (Actual)
Dates: Start 2024-05-13 (Actual); Primary Completion 2024-09-03 (Actual); Study Completion 2024-09-03 (Actual)

PRIMARY OUTCOMES:
Demonstrate the Therapeutic Equivalence & Safety of the Investigational Product | Baseline to Week 12
  Percent change in the inflammatory (papules and pustules) and the non-inflammatory (open and closed comedones) lesion counts.

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Yantovskiy, Study Director — Taro Pharmaceuticals, Inc.
Locations (1):
- Taro Pharmaceuticals USA Inc., Hawthorne, New York, United States

IPD SHARING:
Plan to Share IPD: No